CLINICAL TRIAL: NCT00089518
Title: A Phase III, Randomized, Placebo-Controlled, Double-Blind Trial of an Angiotensin Receptor Blocker (Valsartan) and Highly Active Antiretroviral Therapy (HAART) Versus HAART Alone for the Treatment of HIV-Associated Nephropathy
Brief Title: Optimal Treatment for Kidney Disease in HIV Infected Adults
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACTG A5179
Record Dates: First submitted 2004-08-05; First posted 2004-08-06 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2009-08

CONDITIONS: HIV Infections; Kidney Disease
Keywords: Treatment Experienced
MeSH Terms: conditions — HIV Infections; Kidney Diseases | interventions — Valsartan

INTERVENTIONS:
Drug: Valsartan

SUMMARY:
The angiotensin receptor blocker (ARB) valsartan is a drug commonly used to treat high blood pressure. Valsartan may also help slow down the progression of kidney disease in HIV infected people. The purpose of this study is to compare valsartan and antiretroviral therapy (ART) to ART alone in slowing kidney disease progression in people with HIV.

DETAILED DESCRIPTION:
ART for the treatment of HIV may slow the progression of HIV-associated nephropathy (HIVAN) to end-stage renal disease (ESRD); nevertheless, it is predicted that many HIV infected patients on ART will reach ESRD by the next decade. Medications that affect the renin-angiotensin system, such as the ARB valsartan, may be useful in treating HIVAN. In a small study of HIV infected patients with HIVAN treated with the angiotensin-converting enzyme inhibitor (ACEI) fosinopril, kidney function was stable in patients who took the ACEI, but function decreased in patients who did not. These data are promising, and suggest that an ARB like valsartan may also slow the progression of HIVAN and improve patients' prognosis. This study will compare valsartan and ART to ART alone in slowing kidney disease progression in people with HIV.

This study will last 96 weeks. All participants will continue taking their current ART regimen during the study and will be randomly assigned to one of two arms: Arm 1 will receive valsartan daily, while Arm 2 will receive placebo daily. Doses of drug or placebo may be adjusted during the first 8 weeks based on blood pressure readings taken during the study. In addition, if patients are on other antihypertensive drugs, dosage adjustments may be necessary for those drugs during the study. No ART or antihypertensive drugs other than valsartan will be provided by the study. Study visits will occur every week until Week 8, then every 8 weeks until the end of the study at Week 96. Study visits will include physical examination, medication assessment, and blood pressure readings. In addition, blood collection will occur at entry, Weeks 2, 4, 6, and 8, and every 8 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* Evidence of HIV-associated nephropathy by kidney biopsy performed locally within 24 weeks prior to study entry
* On ART for at least 42 days prior to study entry and willing to continue ART while on study
* Systolic blood pressure (BP) between 91 mm Hg and 170 mm Hg and diastolic BP 105 mm Hg or less within 24 hours of study entry
* Stable kidney function, as indicated by two consecutive calculated creatinine clearance measurements higher than 30 ml/min
* Serum potassium of less than Grade 1 within 7 days prior to study entry
* Willing to follow dose adjustments of non-study antihypertensive drugs if necessary
* Willing to use acceptable forms of contraception

Exclusion Criteria:

* Current treatment with hemodialysis or peritoneal dialysis
* History of kidney transplant
* Condition other than HIVAN contributing to decreased kidney function
* ALT or AST greater than 5 times the upper limit of normal (ULN) within 28 days of study entry
* Total bilirubin greater than 2.5 times ULN within 28 days of study entry. Patients with total bilirubin between 2.5 times and 5 times ULN who are receiving indinavir or atazanavir and do not have cirrhosis or severe liver disease are not excluded.
* Current heart indication for an angiotensin-converting enzyme inhibitor (ACEI) or angiotensin receptor blocker (ARB)
* Use of an ACEI or ARB within 7 days prior to first creatinine clearance measurement obtained for screening or any time between screening and study entry
* Systemic steroid therapy above a replacement level within 28 days of study entry, or possible need for ongoing systemic steroid therapy above replacement level during the study
* Current use of cimetidine
* Use of investigational agents, except when approved by the protocol chairs
* Allergy or sensitivity to valsartan or its formulations
* Blood pressure not measurable by the technique described in the protocol
* Orthostatic drop in systolic BP of 30 mm Hg or more within 24 hours prior to study entry
* Drug or alcohol use that, in the opinion of the investigator, would interfere with the study
* Decreased mental capacity that, in the opinion of the investigator, would interfere with the study
* AIDS-defining opportunistic infection (OI) within 28 days prior to study entry. Patients who are receiving maintenance therapy for OIs and have no evidence of active disease are not excluded.
* Diabetes mellitus for 2 years or longer prior to study entry. Onset of diabetes is defined as the point at which patients began oral hypoglycemics or insulin.
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynda Anne Szczech, MD, MSCE, Study Chair — Division of Nephrology, Department of Medicine, Duke University Medical Center
Locations (10):
- United States (10):
  - Indiana University Hospital, Indianapolis, Indiana
  - Methodist Hospital of Indiana, Indianapolis, Indiana
  - Wishard Hospital, Indianapolis, Indiana
  - Washington University (St. Louis), St Louis, Missouri
  - NYU/Bellevue, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - MetroHealth Medical Center, Cleveland, Ohio
  - Rhode Island Hospital, Providence, Rhode Island
  - Stanley Street Treatment and Resource, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island

REFERENCES:
- [Background] Herman ES, Klotman PE. HIV-associated nephropathy: Epidemiology, pathogenesis, and treatment. Semin Nephrol. 2003 Mar;23(2):200-8. doi: 10.1053/snep.2003.50018. PMID 12704580
- [Background] Kimmel PL, Barisoni L, Kopp JB. Pathogenesis and treatment of HIV-associated renal diseases: lessons from clinical and animal studies, molecular pathologic correlations, and genetic investigations. Ann Intern Med. 2003 Aug 5;139(3):214-26. PMID 12899589
- [Background] Marras D, Bruggeman LA, Gao F, Tanji N, Mansukhani MM, Cara A, Ross MD, Gusella GL, Benson G, D'Agati VD, Hahn BH, Klotman ME, Klotman PE. Replication and compartmentalization of HIV-1 in kidney epithelium of patients with HIV-associated nephropathy. Nat Med. 2002 May;8(5):522-6. doi: 10.1038/nm0502-522. PMID 11984599
- [Background] Wei A, Burns GC, Williams BA, Mohammed NB, Visintainer P, Sivak SL. Long-term renal survival in HIV-associated nephropathy with angiotensin-converting enzyme inhibition. Kidney Int. 2003 Oct;64(4):1462-71. doi: 10.1046/j.1523-1755.2003.00230.x. PMID 12969167